CLINICAL TRIAL: NCT00453115
Title: A Phase II Study of Gemcitabine Plus Oxaliplatin for Patients With Advanced Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine Plus Oxaliplatin in Advanced Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-157
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
Keywords: Non small cell lung cancer; advanced stage IIIB; Stage IV
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental): GemOx
  Interventions: Drug: Oxaliplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Oxaliplatin — oxaliplatin 85mg/m2 iv on D1 and 15, every 4 weeks until disease progression
Drug: Gemcitabine — gemcitabine 1250mg/m2 iv on day 1 and 15, every 4 weeks until disease progression

SUMMARY:
Oxaliplatin is a diaminocyclohexane platinum compound, with a mechanism of action similar to that of cisplatin. Oxaliplatin has a more manageable toxicity profile than cisplatin, with no renal toxicity and a lower incidence of hematological and gastrointestinal toxicities. Gemcitabine and oxaliplatin are both active in NSCLC with no overlapping toxicity. Preclinical studies show a synergistic effect of the gemcitabine-oxaliplatin combination. The combination of gemcitabine-oxaliplatin is attractive in NSCLC patients as it may improve the therapeutic index.

DETAILED DESCRIPTION:
The combination of gemcitabine-oxaliplatin is attractive in NSCLC patients as it may improve the therapeutic index. We are conducting a phase II study to evaluate the response rate and toxicity of the gemcitabine-oxaliplatin combination both given every 4 weeks in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of NSCLC, Stage IV or selected stage IIIB (with positive pleural effusion or separate tumor nodules in the same lobe) according to the American Joint Committee on Cancer (AJCC).
2. No prior chemotherapy.
3. Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
4. No other forms of cancer therapy, such as radiation, immunotherapy for at least 4 weeks before the enrollment in study.
5. Performance status of 0, 1, 2 on the ECOG criteria.
6. At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
7. Estimated life expectancy of at least 12 weeks.
8. Patient compliance that allow adequate follow-up.
9. Adequate organ function including the following:Adequate hematologic function: WBC count ≥ 3,500/uL, absolute neutrophil count (ANC) ≥ 1,500/uL, and platelet count ≥ 100,000/uLAdequate hepatic function: bilirubin ≤ 1.5 x UNL, ALT or AST ≤ 2.5 x UNL.Adequate renal function: creatinine ≤ 1.5mg/dL.
10. Informed consent from patient
11. Males or females at least 18 years old.
12. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study registration.

Exclusion Criteria:

1. MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia
2. Serious concomitant infection including post obstructive pneumonia
3. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
4. Pregnant or nursing women
5. Psychiatric disorder that would preclude compliance.
6. Major surgery other than biopsy within the past two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Response rate | every 12 weeks during until disease progression

SECONDARY OUTCOMES:
To access the toxicity | the first day of the treatment to 30 days after the last dose of study drug
To estimate the time to progression and overall survival | the first day of treatment to the date that disease progression is reported
To evaluate the improvement quality of life | before the first treatment and every cycle d1 until diseas progression
To estimate the overall survival | the first day of the treatment to death date

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-dog, South Korea